CLINICAL TRIAL: NCT00955825
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center, Phase III Study of the Efficacy and Safety of 300 IR Sublingual Immunotherapy (SLIT) Administered as Allergen-based Tablets Once Daily to Adult Patients Suffering From Grass Pollen Rhinoconjunctivitis
Brief Title: Study of Efficacy and Safety of 300 IR Sublingual Immunotherapy (SLIT) Tablets in Adult Patients With Allergic Grass Pollen Rhinoconjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VO61.08 USA
Record Dates: First submitted 2009-08-03; First posted 2009-08-10 (Estimated); Results first posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-04

CONDITIONS: Allergic Rhinitis Due to Grass Pollens
Keywords: allergic rhinoconjunctivitis
MeSH Terms: interventions — Sublingual Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 300 IR (Experimental): 300 IR grass pollen allergen extract tablet
  Interventions: Drug: 300 IR
- Placebo (Placebo Comparator): Pacebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 300 IR — 300 IR grass pollen allergen extract tablet taken daily for approximately 6 months starting 4 months before the grass pollen season and over the grass pollen season
  Other Names: Sublingual immunotherapy tablet
  Arms: 300 IR
Drug: Placebo — Placebo sublingual tablet taken daily for approximately 6 months starting 4 months before the grass pollen season and over the grass pollen season
  Other Names: Sublingual placebo tablet
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the efficacy and safety of 300 IR sublingual tablet of grass pollen allergen extract compared to placebo in adult patient with allergic rhinoconjunctivitis.

DETAILED DESCRIPTION:
Allergy is one of the most common chronic disease in the world currently affecting between 10% and 25% of the general population.

Allergies to pollens characteristically result in seasonal rhinitis symptoms and allergic rhinoconjunctivitis is characterized by sneezing, congestion, rhinorrhea, nasal or palatal itching and itchy, watery, red and swollen eyes.

Even if several drugs effectively manage allergic rhinoconjunctivitis symptoms, immunotherapy is considered more appropriate for patients in whom these symptoms are not optimally controlled with relief medications.

In the study, each of the six rhinoconjunctivitis symptoms (sneezing, runny nose, itchy nose, nasal congestion, itchy eyes, watery eyes) will be evaluated daily and relief medication intake (oral antihistamines, eye drop antihistamine, nasal corticosteroid, oral corticosteroid) reported daily during the grass pollen season.

Efficacy and good safety profile of 300IR SLIT tablet administered once per day for approximately six months (starting 4 months before and over the season) will be demonstrated during the grass pollen season compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Grass pollen-related allergic rhinoconjunctivitis for at least the last two pollen seasons.
2. Positive SPT to grasses
3. Total symptoms score for the previous pollen season more than 12 out of 18.
4. Patients with FEV1 ≥ 80% of the predicted value.

Exclusion Criteria:

1. Positive SPT to other grasses present during the grass pollen season and if endemic to the region
2. Patients with clinically significant confounding symptoms of allergy to other allergens potentially overlapping the grass pollen season
3. Asthma requiring treatment with medications other than beta-2 inhaled agonists.
4. Patients who have received any desensitization treatment for grass pollen in the past 5 years.
5. Ongoing immunotherapy with any other allergen.
6. Patients with any nasal or oral condition that could confound the efficacy or safety assessments
7. Patients with known history of hypersensitivity or intolerance to any of the excipients in the investigational product (such as lactose intolerance).
8. Patients with any past or current clinically significant condition which as judged by the investigator, may affect the patient's participation or the outcome of the study.
9. Patients treated with systemic or inhaled corticosteroids
10. Patients treated or under treatment with beta-blockers, continuous systemic corticotherapy or immunosuppressive drugs.
11. Pregnant, breastfeeding, or sexually active women who are not using a medically accepted contraceptive method as listed above.
12. Patients participating or having participated within 30 days before Screening in any clinical study.
13. Patients who are unlikely to complete the study for any reason, or patients who have to travel for extended periods of time during the grass pollen season which will compromise the data
14. Patients with history of drug or alcohol abuse.
15. Study staff, investigators, sub-investigators, as well as their children or spouses and family members of all study staff should not be enrolled in the study.
16. Patients will not be randomized in this study more than once.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: COX Linda, MD, Principal Investigator — Allergists and Immunologists - Fort Lauderdale - Florida
Locations (19):
- United States (19):
  - Sneeze, wheeze, and Itch Associates, LLC, Normal, Illinois
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Allergy & Asthma Specialists, PSC, Owensboro, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Respiratory Medical Research Institute of Michigan PLC, Ypsilanti, Michigan
  - Clinical Research of the Ozarks, Inc., Columbia, Missouri
  - Midwest Clinical Research LLC, St Louis, Missouri
  - Clinical Research of the Ozarks, Inc, Warrensburg, Missouri
  - Montana Allergy & Asthma Specialists, Billings, Montana
  - Montana Medical Research, Missoula, Montana
  - Creighton University - Allergy & Asthma, Omaha, Nebraska
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Allergy and Asthma Research Group, Eugene, Oregon
  - Baker Allergy, Asthma, & Dermatology Research Center, LLC, Lake Oswego, Oregon
  - Clinical Research Institute of Southern Oregon, P.C., Medford, Oregon
  - Allergy Associates Research, Portland, Oregon
  - Allergy & Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - North West Asthma Allergy Center, Vancouver, Washington

REFERENCES:
- [Result] Cox LS, Casale TB, Nayak AS, Bernstein DI, Creticos PS, Ambroisine L, Melac M, Zeldin RK. Clinical efficacy of 300IR 5-grass pollen sublingual tablet in a US study: the importance of allergen-specific serum IgE. J Allergy Clin Immunol. 2012 Dec;130(6):1327-34.e1. doi: 10.1016/j.jaci.2012.08.032. Epub 2012 Oct 31. PMID 23122534

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient First Visit 22 OCT 2008, Last Patient Last Visit 13 AUG 2009
Groups:
- Placebo: Placebo tablet
Period: Overall Study
Arm/Group | 300 IR | Placebo
Started | 233 | 240
Completed | 207 | 223
Not Completed | 26 | 17
Not completed — Adverse Event | 15 | 2
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Any other reason not above-mentioned | 7 | 9

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) includes all patients who received at least one dose of the investigational product and had at least one Combined Score while on treatment during the pollen period. The FAS was regarded as primary for the efficacy evaluations.
Groups:
- Total: Total of all reporting groups
Arm/Group | 300 IR | Placebo | Total
Number analyzed (Participants) | 210 | 228 | 438
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (11.27) | 37.6 (11.64) | 37.2 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 125 | 234
  Male | 101 | 103 | 204

OUTCOME MEASURES:

1. Primary Outcome: Combined Score (CS)
Description: The daily Combined Score (CS) is a patient specific score taking into account the patient's daily Rhinoconjunctivis Total Symptom Score (RTSS) and daily Rescue Medication Score (RMS), assuming equivalent importance of symptoms and rescue medication scores.
  The RMS (range 0-3) is derived as follows: 0, no rescue medication; 1, use of antihistamine; 2, use of nasal corticosteroid; 3, use of oral corticosteroid. The RTSS (range 0-18) is the sum of the 6 individual rhinoconjunctivitis symptom score (each symptom is scored as follows: 0: no symptoms, 1: mild symptoms, 2: moderate symptoms and 3: severe symptoms).
  The CS (range 0-3) = (RTSS/6 + RMS)/2. The lower the score, the better the outcome.
Time Frame: Pollen period (average of 42.8 days)
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Units on a scale (range: 0 to 3)
Arm/Group | 300 IR | Placebo
Number analyzed (Participants) | 208 | 228
Units on a scale (range: 0 to 3) | 0.32 (0.033) | 0.45 (0.032)
Statistical Analysis 1: Comparison: 300 IR vs Placebo; Test type: Superiority or Other; p = 0.0003, ANCOVA; LS Mean difference vs. Placebo = -0.126, 95% CI [-0.194 to -0.058] — Relative LS Means difference (%) = - 28.24

ADVERSE EVENTS:
Time Frame: 4 months before the pollen period until the end of the pollen period.
Description: A treatment-emergent adverse event (TEAE) is defined as any adverse event that started on or after the first administration of the investigational product.
  Note: Serious Adverse Events and Other Adverse Events are described in the Results Publication.
Arm/Group | 300 IR | Placebo
Serious Adverse Events (participants affected / at risk) | 2/233 | 2/240
Other Adverse Events (participants affected / at risk) | 161/233 | 114/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 300 IR (N=233) | Placebo (N=240)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1
PALATAL DISORDER (Gastrointestinal disorders) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 1
NEUROENDOCRINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 300 IR (N=233) | Placebo (N=240)
NASOPHARYNGITIS (Infections and infestations) | 40 | 42
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 17 | 21
SINUSITIS (Infections and infestations) | 14 | 15
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 54 | 6
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 17 | 15
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 18 | 12
COUGH (Respiratory, thoracic and mediastinal disorders) | 14 | 8
PHARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 12 | 1
ORAL PRURITUS (Gastrointestinal disorders) | 57 | 11
OEDEMA MOUTH (Gastrointestinal disorders) | 22 | 1
PARAESTHESIA ORAL (Gastrointestinal disorders) | 22 | 1
HEADACHE (Nervous system disorders) | 15 | 30
EYE PRURITUS (Eye disorders) | 14 | 7
EAR PRURITUS (Ear and labyrinth disorders) | 31 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No